CLINICAL TRIAL: NCT04084938
Title: Prostatic Artery Embolization vs Transurethral Resection of the Prostate or Open Prostatectomy in Patients With Symptomatic Benign Prostatic Hyperplasia
Brief Title: Artery Embolization vs Operation of Benign Prostate Hyperplasia
Acronym: NORTAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Nils-Einar Kløw, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1231
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Benign Prostatic Hyperplasia; Post-Op Complication; Embolization Therapeutic; Transurethral Resection of Prostate Syndrome
Keywords: Prostate; Embolization; Complication; Operation; Randomization
MeSH Terms: conditions — Prostatic Hyperplasia; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomized study 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate operation (Active Comparator): You will have a surgery to remove the prostate gland. The surgery will be done during general anesthesia. If your prostate gland is small the surgery will be done through a catheter into the penis. If your prostate gland is large the surgery will be through an incision in your lower abdomen.
  Interventions: Procedure: Prostate operation or prostate artery embolization
- Prostate artery embolization (Active Comparator): The embolization is done in the Department of Radiology. There will be placement of a catheter into the artery in one of the groins during local anesthesia. Through this catheter small particles will be injected into the arteries of the prostate gland. When finished, the hole in the artery will be closed.
  Interventions: Procedure: Prostate operation or prostate artery embolization

INTERVENTIONS:
Procedure: Prostate operation or prostate artery embolization — As described above.

SUMMARY:
Aim of the study is to compare prostate artery embolization (PAE) to the established surgical treatment for patient acceptance, morbidity, complications, and the functional outcomes. To compare length of stay, hospital costs and time for recovery. 140 patients will be randomized to PAE or surgery. Patients should suffer from lower urinary tract symptoms (LUTS), be candidates for both treatments and willing to undergo both procedures. Before randomization computed tomography angiography of the pelvic arteries is done to select eligible patients. Magnetic resonance imaging of prostate rules out possible cancer. The PAE is done in the angio suite in the radiology department injecting small particles into the prostate arteries. The surgery is done in the operation room in the urology department according to established procedures. Clinical follow-up include clinical visit after 3 months, 1 and 5 years. Acute as well as long term complications will be recorded.

DETAILED DESCRIPTION:
Background: Prostatic artery embolization (PAE) has recently been described as a promising alternative to surgery for treatment of lower urinary tract symptoms (LUTS) due to an enlarged, benign prostate. The treatment has not been implemented into international guidelines and has only been introduced to few patients in Norway.

Purpose: To compare PAE to the established surgical treatment for patient acceptance, morbidity, complications, and the functional outcomes. To compare length of stay, hospital costs and time for recovery.

Materials and Methods: 140 patients will be randomized to PAE or surgery. Patients should suffer from LUTS, be candidates for both treatments and willing to undergo both procedures. Before randomization computed tomography angiography of the pelvic arteries is done to select eligible patients. Magnetic resonance imaging of prostate rules out possible cancer. The PAE is done in the angio suite in the radiology department injection small particles into the prostate arteries. The surgery is done in the operation room in the urology department according to established procedures. All patients stay in the urology unit after the procedure. Clinical follow-up include clinical visit after 3 months, 1 and 5 years. Acute as well as long term complications will be recorded. The patients fill in the form of quality of life from urologic disease. Urodynamic examination will record functional outcome. Length of stay, procedure costs and recovery time will be recorded.

Importance of the study: Contribute to establishment of new treatment and help to select the right patients for the alternative treatments. Randomized study will give important information to the international community. It is possible to run this study in Norway because it is still in limited use.

ELIGIBILITY:
Inclusion Criteria:

* LUTS from Benign Prostate Hyperplasia (BPH) with moderate and severe IPSS score (IPSS > 8) and QoL = or >3
* and refractory to medical treatment for at least 6 months or the patient is unwilling to accept medical treatment
* or BPH using permanent or intermittent catheterization
* Prostate volume > 50 ml
* Signed informed consent

Exclusion Criteria:

* Urological disorders: evidence of clinically significant prostate cancer [as defined by START criteria] on prostate biopsy (27,28), prostatitis (29,30), detrusor-sphincter dyssynergia or evidence of neurogenic bladder, urethral strictures, bladder neck contracture, bladder stone or bladder cancer
* Renal insufficiency defined as Glomerular Filtration Rate < 30 ml/min/1,73m2
* Known severe reactions to iodine-based contrast or gadolinium-based contrast
* Previous prostate operation
* CT examination reveals no access to the prostate arteries.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life due to urinary symptoms | 3 months
  "Quality of life due to urinary symptoms" QoL = or <3 The scale used: Quality of Life Due to Urinary Symptoms. Scale from 0 to 6, the worse is 6. The patient question: If you were to spend the rest of Your life With Your urinary condition just the way it is now, how would you feel about that?
Number of patients with Prostate Artery Embolization that did not have prostate operation | 12 months
  The investigators will record the number of patients that did not have prostate surgery after Prostate Artery Embolization. After 3 months the patients will be offered operation when Quality of Life Due to Urinary Symptoms is 4-6 on the scale from 0-6 ie. the patients report unsatisfied (4), unhappy (5) or terrible (6).

SECONDARY OUTCOMES:
Number of patients with postoperative complications | 3 months
  Postoperative complications will be recorded according to the Clavien-Dindo classification system. Complication will be recorded during hospital stay, at the follow-up after 3 months and at any intermediate points reported by the patients
Hospital stay | 3 months
  Length of stay including before and after the intervention
Symptoms | 3 months, 1 year, 5 years
  Change in IPSS. The patients fill in the form International Prostate Symptom Score (IPSS) before and after treatment. Seven questions are scored from 0 to 5, 5 is the worst outcome. Total score from 0 - 35. 1-7 is mild symptoms, 8-19 is moderate symptoms, 20-35 is severe symptoms.

OTHER OUTCOMES:
Need for catheters | 3 and 12 months
  Number of patients using permanent and intermittent catheters at follow-up will be recorded
Erectile function | 3 and 12 months
  Change in erectile function will be recoded using the International Index of Erectile Function (IIEF-5) questionnaire. The patients fill in the form before and after treatment. There are 5 questions which score 1-5, 5 is the best. Total score from 5-25.
Ejaculation | 3 and 12 months
  Change in ejaculation will be recorded using the Male Sexual Questionnaire short form for assessing ejaculation. There are 4 questions with 5-6 possible outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Einar Kløw, MD, PHD, Principal Investigator — Department of Radiology, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Aker, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No